CLINICAL TRIAL: NCT06902012
Title: A Prospective, Single - Arm Clinical Study on the Safety and Efficacy of Early Second Infusion of CD19 CAR - T Based on ctDNA Monitoring in the Treatment of Relapsed/Refractory Large B - Cell Lymphoma
Brief Title: Safety and Efficacy of Early Second Infusion of Axi-cel Based on ctDNA for R/R Large B - Cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-343-01
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-02

CONDITIONS: Relapsed/Refractory Diffuse Large B-cell Lymphoma
Keywords: CAR-T; LYMPHOMA; SENCOND INFUSION
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm Group (Experimental): All participants receive early second CAR-T infusion based on ctDNA monitoring.
  Interventions: Drug: Infusion of Axicabtagene Ciloleucel

INTERVENTIONS:
Drug: Infusion of Axicabtagene Ciloleucel — Drug: Axicabtagene Ciloleucel (CD19 CAR-T cells), 2×106 cells/kg, IV infusion at Day 0 and 30-90 days post-first infusion.
  Drug: Cyclophosphamide (500 mg/m²) + Fludarabine (30 mg/m²), IV on Days -5, -4, -3.
  Procedure: ctDNA monitoring via liquid biopsy at pre-lymphodepletion and Months 1, 2, 3, 6, 9, 12 post-infusion.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of early secondary infusion of CD19 CAR T-cell therapy in adults with relapsed/refractory diffuse large B-cell lymphoma (DLBCL), guided by ctDNA monitoring. The main questions it aims to answer are:

1. Efficacy: Does early secondary CAR-T infusion improve the 3-month complete remission (CR) rate and long-term survival outcomes (e.g., 1-year PFS, OS)?
2. Safety: What are the adverse events associated with secondary CAR-T infusion, such as cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity (ICANS), and infections?

This is a single-arm, single-center, prospective study. All participants will receive:

* Leukapheresis to collect T cells for CAR-T manufacturing.
* Preconditioning chemotherapy (fludarabine and cyclophosphamide) to prepare the body for CAR-T infusion.
* Two CD19 CAR-T infusions: The first infusion (2×10⁶ cells/kg) followed by a second infusion (same dose) if ctDNA remains positive when PET/CT shows CR or PET/CT shows PR within 60 days post-first infusion.

Participants will undergo:

* Frequent hospital monitoring for ≥14 days post-infusion to manage potential toxicities.
* Regular follow-ups (e.g., blood tests, ctDNA analysis, PET/CT scans) at scheduled intervals up to 12 months.
* Continuous safety assessments, including CRS grading, neurological evaluations, and infection monitoring.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the efficacy and safety of early secondary infusion of CD19 CAR T-cell therapy in adults with relapsed/refractory diffuse large B-cell lymphoma (DLBCL), guided by ctDNA monitoring. The main questions it aims to answer are:

1. Efficacy: Does early secondary CAR-T infusion improve the 3-month complete remission (CR) rate and long-term survival outcomes (e.g., 1-year PFS, OS)?
2. Safety: What are the adverse events associated with secondary CAR-T infusion, such as cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity (ICANS), and infections?

This is a single-arm, single-center, prospective study. Researchers will enroll 15 eligible participants who have failed prior therapies. All participants will receive:

* Leukapheresis to collect T cells for CAR-T manufacturing.
* Preconditioning chemotherapy (fludarabine and cyclophosphamide) to prepare the body for CAR-T infusion.
* Two CD19 CAR-T infusions: The first infusion (2×10⁶ cells/kg) followed by a second infusion (same dose) if ctDNA remains positive or PET/CT shows incomplete response within 60 days post-first infusion.

Participants will undergo:

* Frequent hospital monitoring for ≥14 days post-infusion to manage potential toxicities.
* Regular follow-ups (e.g., blood tests, ctDNA analysis, PET/CT scans) at scheduled intervals up to 12 months.
* Continuous safety assessments, including CRS grading, neurological evaluations, and infection monitoring.

Key outcomes include 3-month CR rate, objective response rate (ORR), progression-free survival (PFS), overall survival (OS), and incidence of severe adverse events. This trial aims to optimize CAR-T therapy by leveraging ctDNA-guided early intervention to enhance long-term remission in high-risk DLBCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, regardless of gender.
2. Life expectancy >12 weeks.
3. ECOG performance status 0-2.
4. Histologically or cytologically confirmed B-cell non-Hodgkin lymphoma per WHO 2016 classification, including:

   Diffuse large B-cell lymphoma (DLBCL) Primary mediastinal large B-cell lymphoma (PMBCL) Transformed follicular lymphoma (TFL) High-grade B-cell lymphoma (HGBCL).
5. Relapsed/refractory disease, defined as:

   ≥1 prior relapse, Failure to achieve partial response (PR) after 2-3 cycles of first-line therapy, Failure to achieve complete response (CR) after 4-6 cycles of first-line therapy, Primary refractory disease, Secondary refractory disease, Disease progression following last line of therapy.
6. Adequate venous access for leukapheresis, with:

   Hemoglobin ≥80 g/L, Absolute neutrophil count ≥1.0 ×10⁹/L, Platelet count ≥75 ×10⁹/L, OR parameters not meeting above thresholds but deemed acceptable for mononuclear cell collection per investigator's judgment.
7. ≥1 measurable lesion per Lugano 2014 response criteria.
8. Organ function requirements:

   Renal: Serum creatinine ≤2×ULN OR creatinine clearance ≥40 mL/min (Cockcroft-Gault formula).

   Cardiopulmonary:

   Left ventricular ejection fraction (LVEF) >50%, Baseline oxygen saturation >92% on room air.

   Hepatic:

   Total bilirubin ≤2×ULN (≤5×ULN in Gilbert syndrome), ALT/AST ≤3×ULN (≤5×ULN in patients with hepatic involvement).
9. Negative serum pregnancy test for women of childbearing potential (WOCBP). Postmenopausal (≥2 years since last menses) or surgically sterilized women are exempt.
10. Within 60 days post-axi-cel:

Persistent ctDNA(+) or ctDNA(-→+) under CR or PET/CT-confirmed PR

Exclusion Criteria:

1. History of malignancies other than DLBCL, PMBCL, TFL, or HGBCL within 5 years prior to screening, except:

   Adequately treated carcinoma in situ of the cervix, Basal cell or squamous cell carcinoma of the skin, Localized prostate cancer after definitive resection, Ductal carcinoma in situ of the breast after curative surgery, Thyroid cancer after radical treatment.
2. Unstable systemic diseases, including but not limited to:

   Active infections (excluding localized infections), Unstable angina, Cerebrovascular accident or transient ischemic attack (within 6 months prior to screening), Myocardial infarction (within 6 months prior to screening), Congestive heart failure (NYHA Class ≥III), Severe arrhythmia requiring pharmacologic management, Hepatic, renal, or metabolic disorders.
3. Conditions affecting informed consent or protocol compliance:

   Physical or psychological disorders impairing the ability to provide written informed consent, Inability or unwillingness to comply with study requirements.
4. Grade ≥3 cytokine release syndrome (CRS) or immune effector cell-associated neurotoxicity syndrome (ICANS) following prior axi-cel therapy.
5. Active, uncontrolled serious infections.
6. Uncontrolled active comorbidities that preclude study participation.
7. Other conditions deemed by the investigator to confer unacceptable risk or render the patient ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2027-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
complete response rate | 3 months after CAR-T infusion
  the proportion of subjects achieving CR as assessed by the Lugano 2014 criteria (Cheson et al., 2014).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol